CLINICAL TRIAL: NCT01305915
Title: Getting Back on Track: A Single-session Psychoeducational Group Intervention for Women With Breast Cancer Completing Adjuvant Treatment
Brief Title: Getting Back on Track: An Educational Group for Women With Breast Cancer
Acronym: GBOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: The Princess Margaret Cancer Foundation (Other)
Responsible Party: Principal Investigator, Jennifer Jones, Principal Investigator, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 07-0271-CE
Record Dates: First submitted 2011-02-25; First posted 2011-03-01 (Estimated); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
Keywords: single-session group; psychoeducational intervention
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): participant will receive standard print material
- Intervention (Experimental): patient will receive standard print material and a single session group psychoeducational intervention (GBOT)
  Interventions: Behavioral: Getting Back on Track

INTERVENTIONS:
Behavioral: Getting Back on Track — The intervention, entitled Getting Back on Track, is two hours in duration and delivered by a multidisciplinary team representing nursing, radiation therapy, social work, rehabilitation services, and nutrition from the Breast Cancer Clinic at Princess Margaret Hospital. Relying on the content of the Getting Back on Track booklet, clinical experience and the principles of adult education, this team developed scripts for each component of the class.
  Arms: Intervention

SUMMARY:
As the number of women who survive breast cancer continues to grow, more attention is being paid to their quality of life and the disease's long-term effects. The transition from patient to survivor, also termed the "re-entry transition", can be a very difficult and stressful time. A brief psychosocial intervention delivered at this important transition time may address the challenges that women face at re-entry, facilitating greater adaptation and more optimal recovery. The purpose of the proposed RCT is to test the acceptability and effectiveness of a single-session group psychoeducational intervention led by a multi-disciplinary team on adjustment to survivorship. A randomized controlled trial design (RCT) will be used to recruit 440 women attending the breast clinic at Princess Margaret Hospital in Toronto. Participants will be recruited while completing their adjuvant radiotherapy and those who agree to participate will complete the baseline questionnaire package (T0). They then will be randomized to receive either: (1) standard print material (CRL group n=220); or (2) standard print material and a single session group psychoeducational intervention (INT group n=220). Two weeks following randomization, participants in the CRL group will be given the "Getting Back on Track: Life after Treatment" booklet (current standard care), which includes information on the new health care team, physical side-effects, diet and exercise, emotional and social needs and returning to everyday life. Participants in the INT group will receive the same booklet and will also attend a 2- hour psychoeducational group session facilitated by a multidisciplinary team. Participants in both groups will be asked to complete the questionnaire package again at 3 months (post-1) and 6 -months (post-2) following the completion of cancer treatment. Participants in the INV group will also be asked to rate their satisfaction with the class and provide feedback on the content. The proposed intervention will be one of the few clinical interventions designed to address the service gap in helping women to make the transition from patients to survivors by using a single-session psychoeducational group intervention.

ELIGIBILITY:
Inclusion Criteria:

* outpatients attending treatments at PMH
* have a diagnosis of breast cancer;
* have undergone initial treatment for breast cancer;
* are receiving adjuvant radiation therapy as last hospital-based component of treatment;
* are able to speak, read and write English.

Exclusion Criteria:

* metastatic disease
* local recurrence
* cognitive impairment
* if they are an inpatient

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2007-11; Primary Completion 2009-09 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Change in Self Efficacy | Base line, 3 months, 6 months
  Using the Self-Efficacy for Managing Chronic Disease (SEMCDS) questionnaire to measure the change in self efficacy from baseline, to 3 months, and 6 months
Change in Health distress | baseline, 3 months, 6 months
  using the modified Health Distress Scale to assess change in health distress from baseline at 3 months, and at 6 months
Mood State | baseline, 3 months, 6 months
  Profile of Mood States Scale-Short Form (POMS-SF)
Change in Preparedness | baseline, 3 months, 6 months
  Using the Preparedness scale: a 4-item Likert scale questionnaire regarding preparedness adapted from Stanton and Ganz et al (2005), in order to evaluate the change in preparedness from baseline, at 3 months, and at 6 months
Change in Knowledge | baseline, 3 months, 6 months
  measuring changes in knowledge at 3 months and 6 months, compared to baseline using a knowledege questionnaire. This is an 18-item multiple choice questionnaire based on the information booklet and class content will be used to assess knowledge (developed for this study).

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M Jones, PhD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Result] Jones JM, Cheng T, Jackman M, Rodin G, Walton T, Catton P. Self-efficacy, perceived preparedness, and psychological distress in women completing primary treatment for breast cancer. J Psychosoc Oncol. 2010;28(3):269-90. doi: 10.1080/07347331003678352. PMID 20432117